CLINICAL TRIAL: NCT06611605
Title: Effect of Storytelling with Metaphor Toy Used During Venous Blood Collection on Fear and Anxiety Levels in Children: Randomized Controlled Trial
Brief Title: The Effect of Storytelling with Metaphor Toys on Fear and Anxiety Levels in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayla Kaya, Associate Professor, RN, Ph.D, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Akdeniz University TBAEK-602
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: 68 Children Aged 7-10
Keywords: Anxiety; Child; Fear; Nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group = 34 children (Experimental): 34 children aged 7-10 who applied to Akdeniz University Hospital Children's Blood Collection Unit and were subjected to storytelling with metaphor toys
  Interventions: Behavioral: Storytelling with metaphor toys
- Control group = 34 (No Intervention): 34 children aged 7-10 who applied to Akdeniz University Hospital Children's Blood Collection Unit

INTERVENTIONS:
Behavioral: Storytelling with metaphor toys — There is evidence of the effectiveness of various methods such as using different types of balls as tactile stimulation and active distraction methods during the management of pain, anxiety, and fear, watching cartoons, using virtual reality (VR) as a method of distracting attention, and using virtual reality hypnosis (VRH). However, no scientific study has been found on storytelling with a metaphoric toy during venous blood collection.
  Before the children in the intervention group start the blood collection process, the story will be told to the child by the researcher in the waiting room of Akdeniz University Hospital Blood Collection Unit. The child and the parent will be together during the story telling. Expert opinions were received from five academics who completed their doctorate in Child Health and Disease Nursing for the content of the story.
  Arms: Intervention group = 34 children

SUMMARY:
The hospital environment is an unfamiliar environment for children, and unfamiliar people, unknown medical tools and equipment, sounds, and medical procedures in this environment can cause negative emotional states such as fear and anxiety in them. Venous blood collection is one of the most common invasive procedures applied to children who are hospitalized for routine health check-ups or for treatment and care. This procedure can be traumatic enough to create negative emotional states in children and affect them even in their later lives. This study was planned as a randomized controlled experimental study with pre-test-post-test measurements, including intervention (n= 34) and control (n= 34) groups, in order to reduce the fear and anxiety levels of children with the metaphor toy used during venous blood collection. The Child Identification Form, Children Fear Scale, and Children Emotional Manifestation Scale will be used as data collection tools in the study. 68 children between the ages of 7-10 who applied to Akdeniz University Hospital Pediatric Blood Collection Unit will constitute the universe of the research. Data will be collected by face-to-face interview method after receiving institutional permission for the conduct of the research and parental consent. After the final test data collection phase of the research is completed, the obtained data will be analyzed using Statistical Package of Social Science (SPSS) 23.0 software package program. The data evaluation process will be carried out with the support of a statistics expert. It is predicted that the metaphor toy used during the venous blood collection process and storytelling will have lower fear and anxiety levels in the intervention group children compared to the control group children.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study with pre-test-post-test measurements including intervention (n= 34) and control (n= 34) groups in order to reduce fear and anxiety levels in childrens by using a metaphor toy during venous blood collection. The toy to be used in the study was developed by the researchers in order to metaphorize the blood collection process. In the study, the metaphor toy to be used during the blood collection process was used to narrate the bee collecting honey from a flower. In this way, the blood collection process, which can cause fear and anxiety in children, will be metaphorized. The Child Identification Form, Child Fear Scale and Children Emotional Manifestation Scale will be used as data collection tools in the study. 68 children between the ages of 7-10 who applied to Akdeniz University Hospital Pediatric Blood Collection Unit will constitute the universe of the study. Data will be collected by face-to-face interview method after receiving institutional permission for the conduct of the study and parental consent. After the final test data collection phase of the study is completed, the data obtained will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The data evaluation process will be carried out with the support of a statistics expert. It is anticipated that the storytelling with the metaphor toy used during the venous blood collection process will have lower fear and anxiety levels in the intervention group children compared to the control group children.

Intervention Group The research will be implemented in stages. Stage 1: Preliminary Implementation of the Research (First Measurement) A preliminary implementation was conducted with 5 children who met the inclusion criteria of the research in order to evaluate the comprehensibility and applicability of the surveys and storytelling with metaphor toys. After the preliminary implementation, the final version of the application was decided. During the preliminary implementation, a positive change was observed in the emotional states of the children who were applied the intervention after the storytelling with metaphor toys. The children included in the preliminary implementation will not be included in the research sample.

Stage 2: Application After randomization, the pre-test will be applied by the researcher to the children included in the intervention group after obtaining consent from their parents.

The pre-test will be applied to the child who meets the inclusion criteria for the study.

Before the children included in the intervention group proceed to the blood collection process, the story will be told to the child by the researcher in the waiting room of the Akdeniz University Hospital Blood Collection Unit through a metaphor toy. The child and the parent will be together during the story telling. The story presented below will be told to the child in the blood collection unit. Expert opinions were obtained from five academics who completed their doctoral education in the field of Child Health and Disease Nursing for the content of the story.

Stage 3: Post-Test Application (Second Measurement) and Evaluation The post-test (Second Measurement) application will be performed by the researcher immediately after the venous blood collection process is completed.

After the post-test data collection phase of the study is completed, the data obtained will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The data evaluation process will be carried out with the support of a statistics expert.

Control group

* After the informed consent of the parent of the child included in the control group after randomization, the pre-test (First measurement) will be applied by the researcher.
* No application will be made to the children included in the control group.
* The post-test (Second Measurement) will be applied by the researcher immediately after the venous blood collection process is completed.

Data Collection Tools Child Fear Scale (CFS): The Child Fear Scale is used to measure the child fear level. The CFS is a scale that evaluates from 0 to 4, consisting of five drawn facial expressions ranging from a neutral expression (0 = no anxiety) to a frightened face (4 = severe anxiety) and is intended for children aged 5-10. The Turkish validity and reliability study was conducted by Gerçeker et al. in 2018, and this scale can be applied to measure fear before and during the procedure. Permission for use of the scale will be obtained from the responsible author.

Children Emotional Manifestation Scale (CEMS): CEMS was developed by Li Lopez in 2005 to provide nurses with a simple, objective, and consistent method for observing children emotional behaviors during stressful medical procedures. The Cronbach alpha value of the scale was stated as 0.92. Validity and reliability are the most important features that measurement tools should have. Scale adaptation studies include evaluating the reliability and validity of a scale developed in different cultures, testing it in another language and culture, and making it ready for use. The Turkish validity and reliability study of this measurement tool was conducted by Cimke and Bayat in 2021. The Cronbach alpha value of the scale was stated as 0.94. The CEMS consists of 5 sections (Facial Expressions, Sounds, Activity, Interaction, and Cooperation) consisting of emotional behaviors based on observations. In each section, the child receives a score between 1-5. The total score that can be obtained from the scale is between 5 and 25. As the scores obtained from the scale increase, negative emotional indicators increase in direct proportion.

Measurement and evaluation of the effect: In collecting the research data, the Child Identification Form, the Child Fear Scale, and the Children Emotional Manifestation Scale will be used for children. The same measurement tools will be used in collecting the pre-test and post-test data. The intervention will be applied to the children in the intervention group included in the research after the necessary verbal and written permissions are obtained from their parents. No intervention will be applied to the control group. It is planned to apply two measurements, a pre-test and a post-test, to the children in the intervention and control groups. After the completion of the post-test data collection phase of the research, the data obtained will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The data evaluation process will be carried out with the support of a statistics expert.

Randomization: There are 2 groups in the study, 1 intervention group and 1 control group. Simple blind randomization will be performed. Randomization will be performed in the study using the closed envelope method. 34 pieces of paper with intervention 1 and 34 pieces of control written on them will be placed in a closed envelope. A nurse in the blood collection unit will be asked to select a paper from the envelope, independent of the study. Accordingly, the child who accepts to participate in the study will be assigned to the intervention or control group.

Blinding (masking): In order to ensure blinding in the assignment of the sample to the intervention and control groups, children coming to the blood collection unit will be randomly assigned to groups. Since the children assigned to the groups do not know the intervention of the child in the other group except themselves, the sample group will be blinded. In addition, blinding in as many ways as possible is important for the quality and internal validity of the randomized controlled experimental study. In this direction, during the data analysis phase, the database will be created by an expert independent of the research. In order to minimize the risk of bias in the created database, the intervention group will be coded as ''1'' and the control group as ''2'' in the SPSS 23.0 program. The expert from whom statistical support is received will not be informed about the groups.

ELIGIBILITY:
Inclusion Criteria:

* A child between the ages of 7-10 who applied to the Blood Collection Department at Akdeniz University Hospital
* A child whose blood has not been drawn in the last year
* No vision or hearing problems
* No mental or neurological disabilities
* Able to speak and understand Turkish

Exclusion Criteria:

* Wanting to leave the study
* Not accepting the final test application

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Fear level | Change from Baseline (immediately before venous blood collection), immediately after blood collection
  The level of fear will be evaluated among the outcome criteria. The level of fear will be measured with the Child Fear Scale (CFS). The lowest score for CFS is 0 and the highest score is 4. A low score on this scale, which is specific to children, indicates low fear.
Anxiety level | Time Frame: Change from Baseline (immediately before venous blood collection), immediately after blood collection
  The level of anxiety will be evaluated among the outcome criteria. The level of anxiety will be measured with the Children Emotional Manifestation Scale (CEMS). The lowest score for CEMS is 5 and the highest score is 25. A low score on this scale, which is specific to children, indicates low anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Kaya Principal Investigator, Assoc. Prof., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If he/she wishes, he/she can be contacted after the broadcast stage.

REFERENCES:
- [Background] Gerçeker, G. Ö., Ayar, D., Özdemir, Z. & Bektaş, M. (2018). Gaining of Children's State Anxiety and Children's Fear Scale to Turkish Language. E-Journal of Dokuz Eylul University Nursing Faculty, 11(1), 9-13.
- [Background] Li HC, Lopez V. Children's Emotional Manifestation Scale: development and testing. J Clin Nurs. 2005 Feb;14(2):223-9. doi: 10.1111/j.1365-2702.2004.01031.x. PMID 15669931
- [Background] Cimke S, Bayat M. Psychometric Testing of the Turkish Version of Children's Emotional Manifestation Scale. J Pediatr Nurs. 2021 May-Jun;58:60-64. doi: 10.1016/j.pedn.2020.11.008. Epub 2020 Dec 16. PMID 33340936
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301